CLINICAL TRIAL: NCT07092631
Title: Anastomotic Leakage in Colorectal Cancer Surgery in Syria: Risk Factors and Improvements Following Guideline Implementation - A Retrospective Cohort Study
Brief Title: Anastomotic Leakage in Colorectal Cancer Surgery in Syria
Status: Completed | Type: Observational
Sponsor: Elie Bitar (Other)
Collaborators: Syrian Private University (Other); Damascus Hospital (Other)
Responsible Party: Sponsor-Investigator, Elie Bitar, Elie Wadie Bitar MD, Faculty of Medicine, Syrian Private University, Damascus, Syria., Syrian Private University
Organization: Syrian Private University (Other)
Other Study IDs: IRB number 1497/436
Record Dates: First submitted 2025-07-22; First posted 2025-07-30 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Anastomotic Leakage in Colon Surgery; Anastomotic Leak Rectum; Anastomotic Leak Large Intestine
Keywords: general surgery; Syria; leakage; colorectal cancer; rectum; guidelines implementation.
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The First Cohort: Pre-guideline cohort - patients treated before the implementation of the updated hospital guidelines (January 2016 - March 2024).
- The follow-up cohort: Post-guideline cohort - patients treated after the implementation of the updated guidelines (April 2024 - October 2025).

SUMMARY:
Anastomotic leakage is a serious complication of colorectal cancer surgery, particularly in resource-limited and conflict-affected settings. This retrospective cohort study conducted at Damascus Hospital, Syria, evaluated patient and procedure related risk factors for anastomotic leakage following elective sigmoid colon and rectal resections. An initial cohort (January 2016-March 2024) identified modifiable risk factors that informed updates to institutional preoperative and perioperative guidelines. A follow-up cohort (April 2024-October 2025) was subsequently analyzed to assess outcomes after guideline implementation. The study demonstrates that targeted optimization, especially correction of hypoalbuminemia and improved perioperative management was associated with reduced anastomotic leakage and postoperative mortality, highlighting the value of context-specific, evidence-based guideline changes in low-resource surgical settings.

DETAILED DESCRIPTION:
Anastomotic leakage (AL) remains one of the most severe complications following colorectal cancer surgery, leading to substantial morbidity, prolonged hospitalization, increased healthcare costs, and elevated postoperative mortality. The risk and impact of AL are particularly pronounced in low-resource and conflict-affected settings, where limitations in infrastructure, surgical equipment, and perioperative monitoring restrict both prevention and timely management. Despite extensive literature from high-income countries, data from war-affected regions such as Syria remain scarce.

This retrospective cohort study was conducted at the Department of General Surgery, Damascus Hospital, Syria, to identify risk factors associated with AL after elective sigmoid colon and rectal resections for colorectal adenocarcinoma and to evaluate outcomes following the implementation of revised institutional guidelines. The study comprised two sequential cohorts. The first cohort included patients operated on between January 2016 and March 2024 and served to identify patient and procedure related risk factors for AL. Findings from this initial analysis prompted revisions to local preoperative preparation and perioperative management protocols, with particular emphasis on nutritional optimization, correction of hypoalbuminemia, cautious use of perioperative blood transfusion, and intensified postoperative monitoring for high-risk patients.

A follow-up cohort was subsequently analyzed, including patients treated between April 2024 and October 2025 after implementation of the updated guidelines. Outcomes in this cohort were compared with those of the initial cohort to assess the clinical impact of the protocol changes. The primary outcome was the occurrence of anastomotic leakage, defined according to the International Study Group of Rectal Cancer (ISREC) criteria. Secondary outcomes included postoperative complications, perioperative blood transfusion, intensive care unit admission, and postoperative mortality.

All included patients underwent elective resection of the sigmoid colon or rectum for histologically confirmed colorectal adenocarcinoma. Emergency cases, non-neoplastic indications, and incomplete records were excluded. Surgical procedures were classified according to operative approach, anastomotic technique, anastomotic location, and use of diverting ileostomy. Data were retrospectively extracted from medical records and operative notes and verified through structured follow-up when available.

By comparing outcomes before and after guideline implementation, this study aims to demonstrate how locally driven, evidence-based modifications to perioperative care can reduce anastomotic leakage and improve surgical outcomes, even in settings constrained by prolonged conflict and limited resources.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent colorectal cancer surgery for tumor-related indications.

Exclusion Criteria:

* Emergency cases
* Non-tumor related colorectal surgeries

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: from the General Surgery Department of Damascus hospital, Damascus, Syria.
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2016-01-04 (Actual); Primary Completion 2025-10-08 (Actual); Study Completion 2025-10-20 (Actual)

PRIMARY OUTCOMES:
Correlation between preoperative serum albumin level and incidence of anastomotic leakage following colorectal cancer surgery | Within 30 days post-surgery
  Preoperative serum albumin concentration measured in g/dL using routine hospital laboratory biochemical analysis will be correlated with the incidence of anastomotic leakage. Anastomotic leakage will be assessed as a binary outcome (yes/no) based on clinical findings, radiological imaging (contrast-enhanced CT), and/or intraoperative confirmation within the postoperative follow-up period.

CONTACTS AND LOCATIONS:
Locations (1):
- Syrian Private University, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Anastomotic Leakage in Syria- first cohort (2024-07-20): https://cdn.clinicaltrials.gov/large-docs/31/NCT07092631/Prot_SAP_001.pdf
  • Study Protocol: Follow-Up Cohort on Anastomotic Leakage (2025-11-16): https://cdn.clinicaltrials.gov/large-docs/31/NCT07092631/Prot_002.pdf